CLINICAL TRIAL: NCT04072770
Title: Bioavailability of Protein and Amino Acids of Pea Protein Isolate in Healthy Volunteers
Acronym: Qualipois
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Qualipois
Record Dates: First submitted 2019-07-16; First posted 2019-08-28 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Proteins
Keywords: Pea protein; Casein; Amino acid bioavailability; Protein digestibility; Isotopic tracers
MeSH Terms: interventions — Caseins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pea (Experimental): Mashed potatoes meal containing pea protein isolate intrinsically labelled with 15N and 2H
  Interventions: Dietary Supplement: Pea
- Casein (Active Comparator): Mashed potatoes meal containing casein isolate intrinsically labelled with 15N and 2H
  Interventions: Dietary Supplement: Casein

INTERVENTIONS:
Dietary Supplement: Pea — Proteins are intrinsically enriched with 15N and 2H. There are incorporated into mashed potatoes and the test meal is formulated to supply 30 g of pea protein per volunteer.
  Arms: Pea
Dietary Supplement: Casein — Proteins are intrinsically enriched with 15N and 2H. There are incorporated into mashed potatoes and the test meal is formulated to supply 30 g of pea protein per volunteer.
  Arms: Casein

SUMMARY:
The study aims to determine in healthy subjects the bioavailability of protein and amino acids of pea protein isolate and casein isolate. For this purpose, the investigators will compare two methods:

1. the standard method consisting in measuring the ileal digestibility using ileal tubes,
2. an alternative method that has been proposed by an Food and Agriculture Organization (FAO) expert group: the dual isotope method.

DETAILED DESCRIPTION:
2 groups of healthy volunteers are recruited (males and females from 18 to 65 y old), BMI from 18 to 30.

Each group tests a protein source (30g) incorporated in a mashed potatoes that is divided in small portions to perform a repeated meal protocol. Protein sources (pea or casein) are intrinsically labeled with 15N and deuterium (2H).

The day before the meal test, the volunteers are equipped with an intestinal tube that migrates until the ileum. On the day of the experiment, the position of the intestinal tube is checked by radiography in order to verify its location at the terminal ileum. A catheter is inserted in the forearm vein for blood sampling. A saline solution containing polyethylene glycol 4000 (PEG-4000, 20 g/L), used as a non-absorbable marker of the intestinal flow, is infused into the ileum in order to calculate the flow rate of the intestinal effluents. After a basal blood and urine sampling, as well as a basal collection of ileal effluents performed for 30 min, subject ingests at t=0 the first biscuit dose. The small meal portions are ingested every 30 min for 4h, to achieve an isotopic plateau. Tracer doses of carbon 13 (13C) amino acids are ingested concomitantly with the meal doses. Non-absorbable marker (inulin) is added to the test meal to correct for incomplete recovery at the ileal level.

The postprandial sampling period lasts for 8 h after the meal ingestion. The intestinal content is continuously collected over ice and pooled every 30 min. Blood is sampled every 30 min for 4 h, and hourly thereafter.Total urine is collected every 2 h.

Measurements:

In the effluents, the investigators measure PEG 4000, nitrogen (N) and 15N, carbon and 13C, amino acids (AA), 15N and 13C in amino acids and the non-absorbable markers of the meal. The investigators calculate the ileal flow rate, the overall real ileal protein digestibility and the real ileal digestibility of individual amino acids.

In the plasma, the investigators measure uremia and 15N in urea, AA and protein to measure the transfer of dietary N in plasma protein pools; 15N, 2H and 13C in individual amino acids too measure the relative bioavailability of 15N/2H amino acids compared to free 13C amino acids.

In the urine, the investigators measure urea and 15N in the urea ammonia to calculate the postprandial deamination losses.

These measurements will allow to determine the protein and amino acid bioavailability from pea protein and compare it with casein, using the classical method implying ileal sampling and intrinsic tracer of dietary protein (15N). Additionally, it will allow to test a less invasive procedure using multiple tracers to assess the amino acid bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* 18<BMI<30
* Healthy
* Insured under the French social security system
* For women: use of birth control
* Signed informed consent

Exclusion Criteria:

* Any dietary allergy
* Latex allergy
* Positive serology to HIV, hepatite C virus antibody, hepatite B virus surface antigen and core antibodies
* Gluten intolerance
* Anemia
* Use of drugs
* High consumption of alcohol
* Hypertension, diabetes, digestive disease, hepatic or renal disease, severe cardiac disease
* Pregnancy
* High sport practicing (>7h/wk)
* Blood donation in the 3 months prior to the study
* Participation in a clinical study in the 3 months prior to the study
* No signed informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of ileal digestibility of pea proteins and casein | -30 minute to 8 hours after the meal
  Total N and 15N will be measured by Elemental Analyzer coupled to an Isotopic Ratio Mass Spectrometer (EA-IRMS) and the percentage of dietary N reaching the terminal ileum will be then determined. This percentage will be corrected by the ileal flow rate which is estimated with measurement of PEG concentration in effluents by a turbidimetric methods. Ileal digestibility of pea proteins and casein (i.e. N digestibility) will be calculated as 100 - corrected dietary N percentage.
Percentage of ileal digestibility of amino acids from pea proteins and casein | -30 minute to 8 hours after the meal
  Amino acid concentrations will be measured by Ultra High Performance Liquid Chromatography (UHPLC) and 15N, 2H and 13C enrichment in individual amino acids will be measured by Gas Chromatography-Combustion-Isotope Ratio Mass Spectrometry (GC-C-IRMS) in order to determine the percentage of dietary individual amino acids reaching the terminal ileum. This percentage will be corrected by the ileal flow rate which is estimated with measurement of PEG concentration in effluents by a turbidimetric methods. Ileal digestibility of pea and casein amino acid will be calculated as 100 - corrected dietary amino acid percentage.
Percentage of net postprandial protein utilization of pea proteins and casein | -30 minute to 8 hours after the meal
  Urea in plasma and urine (by enzymatic methods) will be determined and associated with 15N enrichment values (by EA IRMS) to determine the 15N transfer in plasma and urinary N pools and calculate the net postprandial protein utilization of pea protein and casein.
Postprandial concentration of dietary amino acids in plasma | -30 minute to 8 hours after the meal
  Concentration of individual amino acids (alanine, arginine, asparagine, aspartic acid, cystein, glutamic acid, glutamine, glycine, histidine, isoleucine, leucine, lysine, methionine, proline, phenylalanine, serine, threonine, valine, tryptophan, tyrosine) in plasma will be determined by UHPLC and associated with 15N enrichment values in individual amino acids (by GC C IRMS) to determined the concentration of dietary amino acids in plasma that comes from pea proteins and casein.
Postprandial concentration of glucose in plasma | -30 minute to 8 hours after the meal
  Concentration of glucose (by enzymatic assay) will be determined in plasma.
Postprandial concentration of insulin in plasma | -30 minute to 8 hours after the meal
  Concentration of insulin (by ELISA) will be determined in plasma.

SECONDARY OUTCOMES:
Validation of the dual isotope method to assess the bioavailability of individual amino acids | -30 minute to 8 hours after the meal
  Measurements of 15N, 2H and 13C amino acids in the plasma by GC-C-IRMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur Volontaires (CRV), Bobigny, Île-de-France Region, France

REFERENCES:
- [Derived] Guillin FM, Gaudichon C, Guerin-Deremaux L, Lefranc-Millot C, Airinei G, Khodorova N, Benamouzig R, Pomport PH, Martin J, Calvez J. Values for the Digestibility of Pea Protein Isolate or Casein Amino Acids Determined using the Dual Isotope Method Are Not Similar to Those Derived with the Standard Ileal Balance Method in Healthy Volunteers. J Nutr. 2024 Feb;154(2):516-525. doi: 10.1016/j.tjnut.2023.12.039. Epub 2023 Dec 29. PMID 38160805
- [Derived] Guillin FM, Gaudichon C, Guerin-Deremaux L, Lefranc-Millot C, Airinei G, Khodorova N, Benamouzig R, Pomport PH, Martin J, Calvez J. Real ileal amino acid digestibility of pea protein compared to casein in healthy humans: a randomized trial. Am J Clin Nutr. 2022 Feb 9;115(2):353-363. doi: 10.1093/ajcn/nqab354. PMID 34665230